CLINICAL TRIAL: NCT02938052
Title: Developing a Positive Psychology Intervention to Promote Health Behaviors in Heart Failure: proof-of Concept Trial
Brief Title: Researching Emotions And Cardiac Health (REACH): Phase II
Acronym: REACH II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Christopher Celano, Assistant in Psychiatry, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016P001443; 1K23HL123607-01A1 (NIH)
Record Dates: First submitted 2016-10-14; First posted 2016-10-19 (Estimated); Results first posted 2018-09-19 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Congestive Heart Failure; Emotions; Patient Compliance
Keywords: Heart Failure; Positive Psychology; Adherence to Health Behaviors
MeSH Terms: conditions — Heart Failure; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention Arm (Experimental): Participants will all undergo a 10-week PP-based health behavior intervention and adherence measurements (baseline and Week 10).
  The participants will receive an ActiGraph accelerometer. They will be asked to begin wearing the accelerometer after their initial visit. Participants will wear the ActiGraph for 7 days at baseline and again at 10 weeks.
  Interventions: Behavioral: PP-based health behavior intervention

INTERVENTIONS:
Behavioral: PP-based health behavior intervention — The positive psychology exercises include 3 modules: Gratitude-based activities, Strength-based activities, and Meaning-based activities. The goal setting exercises include 3 modules: Physical activity, Heart-healthy diet, and Medication adherence.

SUMMARY:
The focus of this study is to examine the feasibility, acceptability, and preliminary impact of our customized positive psychology (PP)-based health behavior intervention in a group of patients with mild to moderate heart failure (HF).

DETAILED DESCRIPTION:
The investigators are proposing a study that will specifically and innovatively focus on the development of a novel positive psychology intervention that is adapted for patients with HF. The MGH inpatient units and MGH Heart Center outpatients will serve as the source of subjects for the study, with patients who have a diagnosis of HF serving as potential subjects. The investigators will enroll 10 HF patients, who will take part in an 10-week PP-based health behavior intervention.

In this project, the investigators hope to do the following:

1. Test an 10-week, telephone-delivered health behavior intervention utilizing PP exercises and systematic goal-setting in a brief, non-randomized, proof-of-concept trial (N=10).
2. Determine whether this initial intervention is feasible in a small cohort of HF patients.
3. Explore potential benefits of the intervention on outcomes of interest (e.g., optimism, positive affect).

Baseline information about enrolled participants will be obtained from the patients, care providers, and the electronic medical record as required for characterization of our population. This information will include data regarding medical history (history of prior acute coronary syndrome, coronary artery bypass graft, congestive HF, hypertension, diabetes mellitus, hyperlipidemia, and current smoking), current medical variables (renal function, left ventricular ejection fraction, NYHA class), medications, and sociodemographic data (age, gender, race/ethnicity, living alone).

Participants will under go an initial visit during which they will meet with study staff in person (or if preferred over the phone).

• They will fill out baseline questionnaires, and be provided a treatment manual with weekly exercises, along with a copy of Learning to Live with Heart Failure. The PP and goal-setting portions of the intervention will be introduced, and the first exercise will be assigned. Finally, participants will be provided an ActiGraph accelerometer to wear for 7 days, as well as a personal step counter to keep.

Participants will undergo weekly phone sessions for 10 weeks.

* For the positive psychology segment the participant will review the previous week's exercise, discuss of the rationale of the next week's exercise, and be assigned the next week's exercise.
* For the goal-setting segment the participant will review the health goal from the prior week, receive education about a health behavior, discuss ways to improve health behaviors, and set a goal for the next week.

Participants will undergo a follow-up phone call at 10 weeks that asks the same questions that were answered during the initial visit, as well as questions about their experience using the ActiGraph.

• At Week 10, participants will wear another ActiGraph for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with NYHA class I, II, or III HF admitted to an MGH inpatient unit or outpatients at the MGH Heart Center. Patients with NYHA class IV HF have ongoing HF symptoms at rest, making it difficult for them to increase physical activity and other health behaviors; therefore, they will not be included. HF diagnosis will be confirmed via chart review and with the patient's treatment team as needed.
* Suboptimal adherence to health behaviors. This will be defined as a total score of ≤15 on three Medical Outcomes Study Specific Adherence Scale (MOS SAS) items regarding diet/exercise/medications. The MOS SAS has been used in multiple prior studies assessing adherence in cardiac patients, including our own studies in this population. This threshold score on the MOS SAS will ensure that all participants will have the potential to improve their health behaviors.

Exclusion Criteria:

* Cognitive deficits impeding a participant's ability to provide informed consent or participate, assessed via a 6-item cognitive test that is sensitive and specific for screening for cognitive impairment in research participants.
* Medical conditions precluding interviews or likely to lead to death within 6 months.
* Inability to speak English, inability to read or write, inability to walk, or lack of a telephone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2017-07-24 (Actual); Study Completion 2017-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Celano, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Celano CM, Freedman ME, Beale EE, Gomez-Bernal F, Huffman JC. A Positive Psychology Intervention to Promote Health Behaviors in Heart Failure: A Proof-of-Concept Trial. J Nerv Ment Dis. 2018 Oct;206(10):800-808. doi: 10.1097/NMD.0000000000000883. PMID 30273277

RESULTS

PARTICIPANT FLOW:
Groups:
- PP-Based Health Behavior Intervention: Participants will all undergo a 10-week PP-based health behavior intervention and adherence measurements (baseline and Week 10).
  The participants will receive an ActiGraph accelerometer. They will be asked to begin wearing the accelerometer after their initial visit. Participants will wear the ActiGraph for 7 days at baseline and again at 10 weeks.
  PP-based health behavior intervention: The positive psychology exercises include 3 modules: Gratitude-based activities, Strength-based activities, and Meaning-based activities. The goal setting exercises include 3 modules: Physical activity, Heart-healthy diet, and Medication adherence.
Period: Overall Study
Arm/Group | PP-Based Health Behavior Intervention
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention Arm: Participants will all undergo a 10-week PP-based health behavior intervention and adherence measurements (baseline and Week 10).
  The participants will receive an ActiGraph accelerometer. They will be asked to begin wearing the accelerometer after their initial visit. Participants will wear the ActiGraph for 7 days at baseline and again at 10 weeks.
  PP-based health behavior intervention: The positive psychology exercises include 3 modules: Gratitude-based activities, Strength-based activities, and Meaning-based activities. The goal setting exercises include 3 modules: Physical activity, Heart-healthy diet, and Medication adherence.
Arm/Group | Intervention Arm
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Positive and Negative Affect Schedule (PANAS) [Mean (Standard Deviation); unit: units on a scale] — The positive affect items on the Positive and Negative Affect Schedule (PANAS), a well-validated scale used in other intervention trials and in patients with HF, will be used to measure positive affect (Range: 10-50). Higher scores indicate higher levels of positive affect. Population: One participant was terminated prior to the completion of baselines as they developed an acute medical illness unrelated to the study.
  units on a scale | 38.70 (3.53)
Life Orientation Test-Revised (LOT-R) [Mean (Standard Deviation); unit: units on a scale] — Life Orientation Test-Revised is a well-validated 6-item instrument used to measure dispositional optimism (Range: 0-24). Higher scores indicate higher levels of optimism. Population: One participant was terminated prior to the completion of baselines as they developed an acute medical illness unrelated to the study.
  units on a scale | 20.90 (2.42)
Hospital Anxiety and Depression Scale (HADS) anxiety subscale [Mean (Standard Deviation); unit: units on a scale] — The Hospital Anxiety and Depression Scale (HADS)-anxiety subscale was be used to measure anxiety. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients (Range: 0-21). Higher scores indicate higher levels of anxiety. Population: One participant was terminated prior to the completion of baselines as they developed an acute medical illness unrelated to the study.
  units on a scale | 4.20 (2.20)
Hospital Anxiety and Depression Scale (HADS) depression subscale [Mean (Standard Deviation); unit: units on a scale] — The Hospital Anxiety and Depression Scale (HADS)-depression subscale was be used to measure depression. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients (Range: 0-21). Higher scores indicate higher levels of depression. Population: One participant was terminated prior to the completion of baselines as they developed an acute medical illness unrelated to the study.
  units on a scale | 1.40 (1.26)
Kansas City Cardiomyopathy Questionnaire (KCCQ) [Mean (Standard Deviation); unit: units on a scale] — The Kansas City Cardiomyopathy Questionnaire is a well-validated questionnaire of health status in HF. The quality of life (QoL) score will be used to measure HF-specific health-related QoL (HRQoL), and the total symptom score will be used as a measure of HF symptoms (QoL score range: 0-100; total symptom score range: 0-100). Higher scores indicate better HF specific health-related QoL and fewer symptoms. Population: One participant was terminated prior to the completion of baselines as they developed an acute medical illness unrelated to the study.
  units on a scale
    HRQoL score | 85.83 (11.82)
    Total Symptom score | 84.06 (15.43)
Medical Outcomes Study Short Form-12 (SF-12) [Mean (Standard Deviation); unit: units on a scale] — The Medical Outcomes Study Short Form-12 (SF-12) will be used to measure quality of life. This is an instrument which has been used in multiple cardiac studies in the past (SF-12 Mental Composite Score and Physical Composite Score Range: 0-100 each). Higher scores represent better health-related quality of life. Population: One participant was terminated prior to the completion of baselines as they developed an acute medical illness unrelated to the study.
  units on a scale
    Physical Health Composite Score | 49.15 (8.05)
    Mental Health Composite Score | 53.57 (6.25)
Medical Outcomes Study Specific Adherence Scale (MOS SAS) [Mean (Standard Deviation); unit: units on a scale] — Three Medical Outcomes Study Specific Adherence Scale (MOS SAS) items assessing medication, diet, and exercise, will be measured individually and as a composite score (Range: 3-18). Higher scores indicate better adherence to health behaviors. Population: One participant was terminated prior to the completion of baselines as they developed an acute medical illness unrelated to the study.
  units on a scale | 12.70 (1.34)
Scored Sodium Questionnaire (SSQ) [Mean (Standard Deviation); unit: units on a scale] — The Scored Sodium Questionnaire (SSQ) is a self-report scale that assesses the frequency with which participants consume a variety of sodium-containing foods, ranging from "Rarely or Never Eaten" to "At Least Once Daily." It is used to calculate daily sodium intake (Range: 0-215). Higher scores indicate higher sodium intake. Population: One participant was terminated prior to the completion of baselines as they developed an acute medical illness unrelated to the study.
  units on a scale | 56.70 (22.38)
Self-Reported Medication Adherence (SRMA) [Mean (Standard Deviation); unit: percentage] — The Self-Reported Medication Adherence (SRMA) asks what percent of the time (in 10% increments) participants took all of their medications as prescribed in the past week and in the past 2 weeks (Range: 0-100). Population: One participant was terminated prior to the completion of baselines as they developed an acute medical illness unrelated to the study.
  percentage | 96.00 (5.16)
Moderate to Vigorous Physical Activity (measured via Actigraph) [Mean (Standard Deviation); unit: minutes/day] — ActiGraph GT3X+ step counters are validated as measures of physical activity and have been used in numerous studies of physical activity in patients with medical illness. In this trial, participants wear the accelerometer for one week at baseline in order to assess average minutes of Moderate to Vigorous Physical Activity (MVPA). Population: 2 participants did not wear the Actigraph and provide adequate data at baseline.
  minutes/day
    number analyzed (Participants) | 9
    (all) | 28.89 (45.29)
Feasibility of Actigraph [Count of Participants; unit: Participants] — Feasibility will be measured by examining the number of participants who use of the Actigraph.
  Participants | 9
Physical Activity [Mean (Standard Deviation); unit: steps/day] — Measured by Actigraph accelerometer, in number of steps per day. Population: Not all participants wore an Actigraph and provided adequate data at baseline.
  steps/day
    number analyzed (Participants) | 9
    (all) | 6435 (6649)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of the PP-based Health Behavior Intervention
Description: Feasibility will be measured by examining the number of completed exercises.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: Exercises Completed
Arm/Group | Intervention Arm
Number analyzed (Participants) | 10
Exercises Completed | 7.8 (2.7)

2. Secondary Outcome: Changes in PANAS Scores
Description: The positive affect items on the Positive and Negative Affect Schedule (PANAS), a well-validated scale used in other intervention trials and in patients with HF, will be used to measure positive affect (Range: 10-50). Change was calculated by subtracting the score at baseline from the score at 10 weeks. Higher scores indicate higher levels of positive affect.
Time Frame: Change in score from Baseline to 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PP-Based Health Behavior Intervention
Number analyzed (Participants) | 9
units on a scale | 2.44 (3.54)

3. Secondary Outcome: Changes in LOT-R Scores
Description: Life Orientation Test-Revised is a well-validated 6-item instrument used to measure dispositional optimism (Range: 0-24). Change was calculated by subtracting the score at baseline from the score at 10 weeks. Higher scores indicate higher levels of optimism.
Time Frame: Change of score from Baseline to 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PP-Based Health Behavior Intervention
Number analyzed (Participants) | 9
units on a scale | 1.56 (1.94)

4. Secondary Outcome: Changes in HADS-Anxiety Subscale Scores
Description: The Hospital Anxiety and Depression Scale (HADS)-anxiety subscale was be used to measure anxiety. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients (Range: 0-21). Change was calculated by subtracting the score at baseline from the score at 10 weeks. Higher scores indicate higher levels of anxiety.
Time Frame: Change in score from Baseline to 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PP-Based Health Behavior Intervention
Number analyzed (Participants) | 9
units on a scale | 2.0 (2.18)

5. Secondary Outcome: Change in HADS-Depression Subscale Scores
Description: The Hospital Anxiety and Depression Scale (HADS)-depression subscale was be used to measure depression. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients (Range: 0-21). Change was calculated by subtracting the score at baseline from the score at 10 weeks. Higher scores indicate worse outcome (i.e. greater levels of depression).
Time Frame: Change in score from Baseline to 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PP-Based Health Behavior Intervention
Number analyzed (Participants) | 9
units on a scale | .11 (1.17)

6. Secondary Outcome: Changes in KCCQ Scores
Description: The Kansas City Cardiomyopathy Questionnaire is a well-validated questionnaire of health status in HF. The full scale will be used to measure HF-specific health-related QoL (HRQoL), and an eight-question subset of the KCCQ will be used as a measure of HF symptoms (QoL score range: 0-100; total symptom score range: 0-100). Change was calculated by subtracting the score at baseline from the score at 10 weeks. Higher QoL scores indicate better HF specific health-related QoL, and higher total symptom scores indicate fewer symptoms.
Time Frame: Change in score from Baseline to 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PP-Based Health Behavior Intervention
Number analyzed (Participants) | 9
units on a scale
  HRQoL score | 5.56 (10.21)
  Total Symptom score | 6.60 (10.44)

7. Secondary Outcome: Changes in SF-12 Scores
Description: The Medical Outcomes Study Short Form-12 (SF-12) will be used to measure quality of life. This is an instrument which has been used in multiple cardiac studies in the past (SF-12 Mental Composite Score and Physical Composite Score Range: 0-100 each). Change was calculated by subtracting the score at baseline from the score at 10 weeks. Higher scores indicate higher level of health related QoL.
Time Frame: Change in score from Baseline to 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PP-Based Health Behavior Intervention
Number analyzed (Participants) | 9
units on a scale
  Physical Health Composite Score | 2.44 (7.38)
  Metal Health Composite Score | 2.17 (6.65)

8. Secondary Outcome: Changes in MOS SAS Scores
Description: Three Medical Outcomes Study Specific Adherence Scale (MOS SAS) items assessing medication, diet, and exercise, will be measured individually and as a composite score (Range: 3-18). Change was calculated by subtracting the score at baseline from the score at 10 weeks. Higher scores indicate better adherence to health behaviors.
Time Frame: Change in score from Baseline to 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PP-Based Health Behavior Intervention
Number analyzed (Participants) | 9
units on a scale | 2.78 (2.33)

9. Secondary Outcome: Changes in Daily Sodium Intake (as Measured With the SSQ)
Description: The Scored Sodium Questionnaire (SSQ) is a self-report scale that assesses the frequency with which participants consume a variety of sodium-containing foods, ranging from "Rarely or Never Eaten" to "At Least Once Daily." It is used to calculate daily sodium intake (Range: 0-215). Change was calculated by subtracting the score at baseline from the score at 10 weeks. Higher scores indicate higher sodium intake.
Time Frame: Change in score from Baseline to 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PP-Based Health Behavior Intervention
Number analyzed (Participants) | 8
units on a scale | 16.31 (18.92)

10. Secondary Outcome: Self-Reported Medication Adherence (SRMA)
Description: The Self-Reported Medication Adherence (SRMA) asks what percent of the time (in 10% increments) participants took all of their medications as prescribed in the past week and in the past 2 weeks (Range: 0-10). Change was calculated by subtracting the score at baseline from the score at 10 weeks.
Time Frame: Change in score from Baseline to 10 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | PP-Based Health Behavior Intervention
Number analyzed (Participants) | 9
percentage of time | .44 (.53)

11. Secondary Outcome: Change in Physical Activity
Description: Measured by Actigraph accelerometer, in number of steps per day.
Time Frame: Baseline and 10 weeks
Population: Not all participants wore the Actigraph and provided adequate data.
Measure: Mean (Standard Deviation); unit: steps/day
Arm/Group | PP-Based Health Behavior Intervention
Number analyzed (Participants) | 8
steps/day | 706 (1616)

12. Secondary Outcome: Change in Moderate to Vigorous Physical Activity (Actigraph)
Description: ActiGraph GT3X+ step counters are validated as measures of physical activity and have been used in numerous studies of physical activity in patients with medical illness. In this trial, participants will wear the accelerometer for one week at baseline and again for one week at 10 weeks to assess the feasibility of doing so and to ensure adequate capture of physical activity. Change was calculated by subtracting the MVPA at baseline from the MVPA at 10 weeks.
Time Frame: Change in MVPA from Baseline to 10 weeks
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | PP-Based Health Behavior Intervention
Number analyzed (Participants) | 8
minutes/day | .15 (9.97)

13. Secondary Outcome: Feasibility of Actigraph
Description: Feasibility will be measured by examining the number of participants who use of the Actigraph.
Time Frame: Baseline and 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | PP-Based Health Behavior Intervention
Number analyzed (Participants) | 10
Participants
  Baseline Actigraph | 9
  10 Week Actigraph | 8

14. Secondary Outcome: Acceptability of the Exercises: Utility Score
Description: Participants will provide ratings of utility after each exercise, measured on a 10-point Likert scale (0-10). Higher scores indicate greater utility of the exercise. Weekly utility ratings were averaged to provide an overall utility score of the exercises.
Time Frame: Weeks 1-10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 10
units on a scale | 7.8 (1.8)

15. Secondary Outcome: Acceptability of the Exercises: Ease Score
Description: Participants will provide ratings of ease after each exercise, measured on a 10-point Likert scale (0-10). Higher scores indicate greater ease of the exercise. Weekly ease ratings were averaged to provide an overall easy score of the exercises.
Time Frame: Weeks 1-10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 10
units on a scale | 7.5 (2.1)

16. Secondary Outcome: Immediate Impact of the Exercises: Optimism Rating
Description: Participants will provide ratings of optimism before and after each exercise, measured on a 10-point Likert scale (0-10). Weekly pre- and post-exercise ratings of optimism were averaged to provide an overall pre- and post-exercise optimism score. Higher scores indicate higher levels of optimism.
Time Frame: Weeks 1-10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PP-Based Health Behavior Intervention
Number analyzed (Participants) | 10
units on a scale
  Pre-Exercise Rating | 8.2 (1.5)
  Post-Exercise Rating | 8.4 (1.3)

17. Secondary Outcome: Immediate Impact of the Exercises: Positive Affect Rating
Description: Participants will provide ratings of positive affect, before and after each exercise, measured on a 10-point Likert scale (0-10). Weekly pre- and post-exercise ratings of happiness were averaged to provide an overall pre- and post-exercise score. Higher scores indicate higher levels of positive affect.
Time Frame: Weeks 1-10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PP-Based Health Behavior Intervention
Number analyzed (Participants) | 10
units on a scale
  Pre-Exercise Rating | 7.8 (1.5)
  Post-Exercise Rating | 8.6 (1.1)

ADVERSE EVENTS:
Time Frame: 1 year and 8 months
Arm/Group | Intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 1/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Arm (N=10)
Unexpected Fall (Injury, poisoning and procedural complications) | 1 (1) — Participant had an unexpected fall 1 week after completing baselines and broke their hip.
Arrhythmia (Cardiac disorders) | 1 (1) — Participant had an arrhythmia while at work and was hospitalized.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Arm (N=10)
Small, unexpected fall (Injury, poisoning and procedural complications) | 1 (1) — Participant reported a small fall while exiting his car post-exercise. No significant injury resulted and participant recovered quickly.

LIMITATIONS AND CAVEATS:
Was performed at a single academic medical center and had a largely White population. It was a small sample size and there was no control condition in this initial trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-28): https://cdn.clinicaltrials.gov/large-docs/52/NCT02938052/Prot_SAP_000.pdf